CLINICAL TRIAL: NCT07319325
Title: Efficacy of an Adaptive, Gamified Digital Therapeutics Intervention for Individuals With Methamphetamine Use Disorder in Community Rehabilitation: A Pragmatic Randomized Controlled Trial
Brief Title: Efficacy of Adaptive, Gamified Digital Therapeutics Intervention for Individuals With Methamphetamine Use Disorder in Community Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JK2025
Record Dates: First submitted 2025-12-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Addiction
Keywords: Digital Therapeutics; Cognitive Bias Modification; Approach Bias Modification; Community Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Digital Therapeutics (DTx) (Experimental): Participants receive access to WonderLab Harbor+ (Adaptive DTx), a smartphone application, for 8 weeks. They are instructed to complete one ICBT session per week (approx. 10 mins) and one Adaptive Approach Bias Modification (A-ApBM) session daily (approx. 3 mins). The app also includes cognitive training games and a rewards system (Contingency Management). This is provided in addition to standard community care.
  Interventions: Device: WonderLab Harbor+ (Adaptive DTx)
- Treatment as Usual (TAU) (Active Comparator): Participants receive standard care provided by the community rehabilitation centers, which consists of counseling sessions (in-person or telephone) delivered by social workers covering stress management, family issues, and craving suppression.
  Interventions: Behavioral: Standard Community Counseling

INTERVENTIONS:
Device: WonderLab Harbor+ (Adaptive DTx) — Participants receive access to a smartphone application for 8 weeks. They are instructed to complete one ICBT session per week (approx. 10 mins) and one Adaptive Approach Bias Modification (A-ApBM) session daily (approx. 3 mins). The app also includes cognitive training games and a rewards system (Contingency Management). This is provided in addition to standard community care.
  Arms: Adaptive Digital Therapeutics (DTx)
Behavioral: Standard Community Counseling — Participants receive standard care provided by the community rehabilitation centers, which consists of counseling sessions (in-person or telephone) delivered by social workers covering stress management, family issues, and craving suppression.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study evaluates the efficacy of a comprehensive, adaptive digital therapeutics (DTx) smartphone application compared to treatment as usual (TAu) for individuals with Methamphetamine Use Disorder (MUD) receiving community-based rehabilitation. The intervention integrates Internet-based Cognitive Behavioral Therapy (ICBT), adaptive Approach Bias Modification (A-ApBM), cognitive training, and contingency management. The primary hypothesis is that the DTx intervention will result in a greater reduction in cue-induced craving compared to standard community care.

DETAILED DESCRIPTION:
Methamphetamine Use Disorder (MUD) lacks effective pharmacotherapies, and traditional psychosocial interventions face scalability challenges in community settings. This pragmatic randomized controlled trial (RCT) aims to assess a smartphone-based digital therapeutic intervention designed to overcome these barriers.

Participants recruited from 12 community rehabilitation centers in Sichuan, China, are randomized 1:1 to either the DTx group or the Treatment as Usual (TAu) group.

The DTx group uses a smartphone application ("WonderLab Harbor+") for 8 weeks as an adjunct to standard care. The app includes:

1. Weekly Internet-based CBT sessions.
2. Daily Adaptive Approach Bias Modification (A-ApBM) training, which dynamically adjusts difficulty based on performance.
3. Gamified cognitive function training.
4. A contingency management system rewarding adherence.

The TAu group receives standard counseling services provided by community social workers. The primary outcome is the change in self-reported cue-induced craving from baseline to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Currently enrolled in a community rehabilitation program.
* Ability to fluently operate a smartphone (Android or iOS).

Exclusion Criteria:

* Presence of a severe mental health condition (e.g., schizophrenia, bipolar I disorder) requiring acute psychiatric care.
* Inability to provide informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Cue-Induced Craving Score | Baseline and 8 Weeks (Post-intervention)
  Self-reported craving elicited by standardized methamphetamine-related images, measured using a Visual Analog Scale (VAS). Scores range from 0 to 100, with higher scores indicating higher craving. The outcome is defined as the change in score from Baseline to Week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Rehabilitation Centers, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon reasonable request to the corresponding author.
Supporting Information: Analytic Code

REFERENCES:
- [Result] Zhang L, Li N, Li Y, Zhang T, Li D, Liu Y, Liu X, Hao W. Preliminary efficacy of a digital therapeutics smartphone application for methamphetamine use disorder: An experimental study. Front Psychiatry. 2022 Oct 19;13:1027695. doi: 10.3389/fpsyt.2022.1027695. eCollection 2022. PMID 36339836
- [Result] Shen D, Jiao J, Zhang L, Liu Y, Liu X, Li Y, Zhang T, Li D, Hao W. Gamified Adaptive Approach Bias Modification in Individuals With Methamphetamine Use History From Communities in Sichuan: Pilot Randomized Controlled Trial. JMIR Serious Games. 2025 Mar 10;13:e56978. doi: 10.2196/56978. PMID 40063843